CLINICAL TRIAL: NCT04213196
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability and Pharmacokinetics of HSK21542 in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of HSK21542 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSK21542-102
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- HSK21542 0.2 μg/kg（15 min) (Experimental): Healthy volunteers 0.2 μg/kg HSK21542
  Interventions: Drug: HSK21542
- HSK21542 0.5 μg/kg (Experimental): Healthy volunteers 0.5 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542
- HSK21542 1 μg/kg （15min) (Experimental): Healthy volunteers 1 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542
- HSK21542 1 μg/kg （2min) (Experimental): Healthy volunteers 1 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542
- HSK21542 0.75 μg/kg (Experimental): Healthy volunteers 0.75 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542
- HSK21542 1.5 μg/kg (Experimental): Healthy volunteers 1.5 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542
- HSK21542 2.25 μg/kg (Experimental): Healthy volunteers 2.25 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542
- HSK21542 3.375 μg/kg (Experimental): Healthy volunteers 3.375 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542
- HSK21542 0.2 μg/kg（2min) (Experimental): Healthy volunteers 0.2 μg/kg HSK21542 or Placebo
  Interventions: Drug: HSK21542

INTERVENTIONS:
Drug: HSK21542 — Intravenous injection 0.2 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 15 min.
  Other Names: HSK21542 0.2 μg/kg
  Arms: HSK21542 0.2 μg/kg（15 min)
Drug: HSK21542 — Intravenous injection 0.5 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 15 min.
  Other Names: HSK21542 0.5 μg/kg
  Arms: HSK21542 0.5 μg/kg
Drug: HSK21542 — Intravenous injection 1 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 15 min.
  Other Names: HSK21542 1 μg/kg
  Arms: HSK21542 1 μg/kg （15min)
Drug: HSK21542 — Intravenous injection 1 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 2 min.
  Other Names: HSK21542 1 μg/kg
  Arms: HSK21542 1 μg/kg （2min)
Drug: HSK21542 — Intravenous injection 0.75 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 15 min.
  Other Names: HSK21542 0.75 μg/kg
  Arms: HSK21542 0.75 μg/kg
Drug: HSK21542 — Intravenous injection 1.5 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 15 min.
  Other Names: HSK21542 1.5 μg/kg
  Arms: HSK21542 1.5 μg/kg
Drug: HSK21542 — Intravenous injection 2.25 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 15 min.
  Other Names: HSK21542 2.25 μg/kg
  Arms: HSK21542 2.25 μg/kg
Drug: HSK21542 — Intravenous injection 3.375 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 15 min.
  Other Names: HSK21542 3.375 μg/kg
  Arms: HSK21542 3.375 μg/kg
Drug: HSK21542 — Intravenous injection 0.2 μg/kg solution (active or placebo, 0.5-1h after standard meal). Complete infusion within 2 min.
  Other Names: HSK21542 0.2 μg/kg
  Arms: HSK21542 0.2 μg/kg（2min)

SUMMARY:
This is a first-in-human, Phase I, single-dose escalation clinical trial conducted in Chinese healthy volunteers. The safety, tolerability, and PK of HSK21542 injection in healthy volunteers will be evaluated using a randomized, double-blind, placebo-controlled trial design

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-45 years old (inclusive) at screening;
2. Male volunteers no less than 50 kg, or female volunteers no less than 45 kg, with body mass index [BMI] in the range of 18.0-27.0 kg/m2 (inclusive) at screening;
3. Healthy volunteers, as assessed by the investigator based on past medical history, comprehensive physical examination, vital signs, and specified tests and examinations.
4. Fully understand the nature, purpose, and potential benefits, inconveniences and risks of the trial. Understand the study procedure and voluntarily provide written informed consent.
5. Able to communicate with the investigator and to follow all requirements of the study, and willing to be admitted into the phase I clinical facility.

Exclusion Criteria:

1. Those who have suffered or are currently suffering from any clinical serious disease such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormality or any other disease or physiological condition that can interfere with the results;
2. Physical examination, vital sign monitoring, ECG examination, chest anteroposterior and lateral radiographs, laboratory examination (including blood routine, urine routine, blood biochemistry, coagulation function, thyroid function, blood pregnancy (only for female subjects) during screening period, and the researcher judged that the abnormality had clinical significance;
3. People with positive hepatitis B surface antigen, positive hepatitis C antibody, positive Treponema pallidum antibody, or positive AIDS virus antibody test;
4. Patients with QTcF>450 ms in ECG examination during screening;
5. Allergic constitution: such as those who are allergic to two or more drugs and foods; Or those who are allergic to any ingredient in this product and auxiliary materials; (Auxiliary materials: glacial acetic acid, sodium acetate, water for injection)
6. Those who cannot tolerate venipuncture and/or have a history of blood and needle sickness;
7. Those who have drunk too much tea, grapefruit, coffee, caffeinated or grapefruit drinks for a long time (more than 8 cups a day, 1 cup=250mL);
8. Those who have a history of alcohol abuse within 3 months before screening, that is, those who drink more than 14 units of alcohol per week (1 unit=12 ounces or 360 mL of beer, 1.5 ounces or 45 mL of spirits with 40% alcohol content, 5 ounces or 150 mL of wine), or those who have positive alcohol breath test;
9. Volunteers with a positive urine nicotine test;
10. Volunteers with drug abuse or dependence, or with a positive urine drugs of abuse test;
11. Those who have used any prescription medicine, over-the-counter medicine, Chinese herbal medicine and health care products within 14 days
12. Blood donation or loss of blood > 450 mL within the past 3 months;
13. Participation in any clinical trials within the past 3 months;
14. Volunteers who plan to become pregnant within the next 6 months;
15. Any other factors judged by the investigator to be unsuitable for participating in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
AE/serious AE | From screening up to 3 weeks
  Adverse event/serious adverse event
Vital signs: Systolic and Diastolic Blood Pressure | From screening up to 3 weeks
  Vital signs (Systolic and Diastolic Blood Pressure) will be collected in healthy volunteers.
Ramsay sedation score | -60 minutes before administration until 24 hours after administration
  Ramsay sedation score will be collected
Visual analog scale (VAS) addiction score | from administration to 24 hours after administration
  VAS addiction score will be collected

SECONDARY OUTCOMES:
Peak concentration (Cmax) | -30 minutes before administration until 24 hours after administration
  Cmax（a measure of the body's exposure to HSK21542）will be calculated in healthy volunteers.
Area under the concentration-time curve（AUC） | -30 minutes before administration until 24 hours after administration
  AUC（a measure of the body's exposure to HSK21542）will be calculated in healthy volunteers.
Tmax | -30 minutes before administration until 24 hours after administration
  time to peak observed
Total clearance | -30 minutes before administration until 24 hours after administration
  Total clearance
Prolactin level | before administration until 24 hours after administration
  Prolactin level will be collected
Antidiuretic hormone level | before administration until 24 hours after administration
  Antidiuretic hormone level will be collected
Urine volume | before administration until 24 hours after administration
  Urine volume will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, PhD, Study Director — The Second Affiliated Hospital of Zhejiang University Medical College; Hong-gang Lou, PhD, Study Director — The Second Affiliated Hospital of Zhejiang University Medical College
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zollner C, Mousa SA, Fischer O, Rittner HL, Shaqura M, Brack A, Shakibaei M, Binder W, Urban F, Stein C, Schafer M. Chronic morphine use does not induce peripheral tolerance in a rat model of inflammatory pain. J Clin Invest. 2008 Mar;118(3):1065-73. doi: 10.1172/JCI25911. PMID 18246198